## Statistical Analysis Plan

**Study Title:** Grant Title: RELAX: A mobile application suite targeting obesity and stress NCT02615171

## Statistical Analysis Plan

Study Title: Grant Title: RELAX: A mobile application suite targeting obesity and stress

We summarized retention, app use, usability, acceptability, and burden using descriptive statistics. For variables that were normally distributed, we described distributions using mean and standard deviation (M[SD]), and for variables that were not normally distributed, we described distributions using median and inter-quartile range (IQR). We compared retention and acceptability by treatment condition using chi-squared tests, or Fisher's exact tests as appropriate. We compared treatment conditions on app usability using a t-test and app burden using a Wilcoxon rank-sum test. We took an intent-to-treat approach to describing weight change. For 2 participants (one in each condition) who became pregnant during the study, we used latest available pre-pregnancy weights (from weeks 2 and 3, respectively). For the three participants who did not provide weight at follow-up, we also used their latest weight from their study scale (weeks 6, 9, and 10, respectively).